CLINICAL TRIAL: NCT00260377
Title: Aspirin Resistance Following Coronary Bypass Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The researcher had left the hospital and the project was stopped
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-03-3107-JL-CTIL
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Ischemic Heart Disease
Keywords: Aspirin treatment; Aspirin resistance; Coronary bypass surgery
MeSH Terms: conditions — Myocardial Ischemia | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Coronary artery bypass surgery

SUMMARY:
Aspirin was proved to be the drug preventing vein grafts from closure and improving clinical outcome after coronary artery bypass surgery. It appears to be effective when being prescribed as early as first 48 hr. after the operation without increasing the incidence of bleeding complications. the exact effective dose is not known.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Coronary artery bypass surgery
* Patients who signed Informed Consent Form

Exclusion Criteria:

* Concomitant valve surgery or carotid surgery or off-pump surgery
* Need for anticoagulation therapy for any reason
* Another antiplatelet medications at least 7 days prior to surgery
* Contra-indication for aspirin treatment
* Thrombocytopenia / thrombocytopathia
* NSAIDs treatment for chronic medical conditions
* Reluctance to participate in the study

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2006-06; Study Completion 2006-12

PRIMARY OUTCOMES:
Ventilation
Inotropic support
Mortality
Perioperative MI
Perioperative stroke
Bleeding / reopen / transfusion
Dysrhythmias

SECONDARY OUTCOMES:
ICU stay
In-hospital stay
Non-fatal cardiac events - MI, recurrence of angina, dysrhythmias
Need for repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lavee, Dr, Principal Investigator — jacob.lavee@sheba.health.gov.il
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel